CLINICAL TRIAL: NCT05478473
Title: Clinical Study of Chidamide Combined With Toripalimab in the Treatment of Advanced Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q31
Record Dates: First submitted 2022-07-27; First posted 2022-07-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with Toripalimab (Experimental)
  Interventions: Drug: Chidamide combined with Toripalimab

INTERVENTIONS:
Drug: Chidamide combined with Toripalimab — chidamide：oral, 30 mg/time, twice weekly; Toripalimab：intravenous drip, 240mg, once every 3 weeks

SUMMARY:
The study was a single-arm study designed to evaluate the efficacy and safety of Chidamide combined with Toripalimab.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years, male or female
* histologically and/or cytologically confirmed melanoma, clinically diagnosed as inoperable stage III-IV
* previous treatment for advanced tumors (including chemotherapy, targeted, anti-vascular drugs, etc.) failure or no standard treatment, and no PD- (L) 1/CTLA-4 drug treatment; if neoadjuvant/adjuvant therapy has received PD- (L) 1/CTLA-4 drug treatment, the total duration of drug treatment should be ≥6 months
* if there is brain metastasis, local treatment must have been received before participating in this study and clinical stability ≥ 3 months
* ECOG score 0-1
* at least one measurable lesion (according to RECISTv1.1 evaluation criteria)
* absolute neutrophil count ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L
* other organ function needs to meet: ① cardiac function needs to meet: left ventricular ejection fraction ≥ 50%, no organic arrhythmia; ② liver function needs to meet: ALT and AST ≤ 2.5 times the upper limit of normal (such as with liver metastasis, ALT and AST ≤ 5 times the upper limit of normal), total bilirubin ≤ 1.5 times the upper limit of normal;③ renal function needs to meet: creatinine ≤ 1.5 times the upper limit of normal; ④ coagulation function: international normalized ratio (International Normalized Ratio,INR) ≤ 1.5 times upper limit of normal; prothrombin time (PT), activated partial thromboplastin time (APTT) ≤ 1.5 times upper limit of normal (unless the subject was receiving anticoagulant therapy and PT and APTT were within the expected range of anticoagulant therapy at screening); ⑤ Thyroid function: thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were within ± 10% of normal values.
* Expected survival time ≥ 3 months
* Voluntarily participate in this clinical trial and sign a written informed consent.
* Previous anti-tumor therapy (chemotherapy, radiotherapy, targeting, traditional Chinese medicine, other immunotherapy) requires eluting for 28 days.
* The adverse effects of previous antitumor therapy were resolved to grade 0-1 before the screening period (as determined by NCI CTCAE 5.0; Except for toxicity, such as hair loss, which the investigator determined did not pose a safety risk to the subject)

Exclusion Criteria:

* no measurable lesions, such as pleural or pericardial exudates, ascites, etc.
* choroidal melanoma
* previous treatment with HDAC inhibitors (including cedaramide, romidepsin, vorinostat, bellistat, panobinostat, etc.)
* history of interstitial lung disease or pneumonia requiring oral or intravenous steroids
* previous vaccination or planned vaccination with live vaccines (seasonal influenza vaccine without live vaccines is allowed), major surgery within 30 days before the first study treatment
* active infection [active bacterial, viral, fungal, mycobacterial, parasitic infections or other infections (excluding fungal infections of the nail bed) within 4 weeks before the screening period, or any major infection event requiring intravenous antibiotic therapy, or targeted antiviral therapy, or hospitalization; Active hepatitis is defined as HBsAg positive with HBV DNA≥500 IU/ml or HCV antibody positive with HCV copy number > the upper limit of normal], or persistent fever within 14 days before screening
* history of immunodeficiency, including positive HIV testing, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation
* uncontrolled cardiovascular disease; history of clinically significant QT prolongation, or screening period > 470 ms for females and > 450 ms for males
* positive baseline pregnancy test in female subjects who are pregnant or lactating or fertile females; or subjects of childbearing age who are unwilling to take effective contraceptive measures for at least 180 days during study participation and after the last dose of study drug
* According to the investigator 's judgment, there are concomitant diseases that seriously jeopardize the subject' s safety or affect the subject 's completion of the study (e.g., severe hypertension ≥ 180/110 mmHg, uncontrolled diabetes, thyroid disease, Hypertriglyceridemia ≥ grade 2, etc.)
* History of definite neurological or psychiatric disorders, including epilepsy or dementia
* Any condition that, in the opinion of the investigator, would make participation in this study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR)as measure of efficacy by RECIST 1.1

SECONDARY OUTCOMES:
Progression Free survival （PFS） | Up to approximately 24 months
  Defined as the time from first dosing (C1D1) to date of first observed progression or death from any cause (whichever comes first)
Overall Survival（OS） | Up to approximately 24 months
  OS as measure of efficacy by RECIST 1.1
Duration of Response(DoR) | Up to approximately 24 months
  DoR as measure of efficacy by RECIST 1.1
Disease control rate（DCR） | Up to approximately 24 months
  Defined as the percentage of patients who have achieved a confirmed response of at least CR or PR or a response of SD
Incidence Rate of each Toxicity (safety and tolerability) | Up to approximately 24 months
  safety and tolerability as measure of efficacy by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China